CLINICAL TRIAL: NCT03515889
Title: A Trial of the Ideal Protein System Versus Low Fat Diet for Weight Loss
Acronym: RENEWAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Ideal Protein (Unknown)
Responsible Party: Principal Investigator, Lydia A. Bazzano, Associate Professor of Epidemiology, Tulane University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-917
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants (n=192) with BMI ≥30 and ≤49 will be randomized to one of two parallel study arms: Group A: Ideal Protein Weight Loss Intervention; Group B: Standard Low-Fat, Low-Calorie, Guideline-based Weight Loss Intervention. Participants will undergo baseline testing, and if eligible, will be randomly assigned to study group, undergo three months of their assigned study intervention, and clinical testing at baseline, 6, and 12 weeks.
Who Masked: Outcomes Assessor
Masking Description: Throughout the study every effort will be made to ensure objective and blinded assessments of outcomes. Although participants will be told of their treatment assignment they will not be provided details about the intervention techniques of the other treatment groups. Focus will instead be maintained on the group to which they are assigned. Staff who obtain and record participant assessments at the clinical assessments will not be informed of the participant's treatment assignment and will not participate in the delivery of the study interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ideal Protein Weight Loss Protocol (Experimental): This arm will follow the Ideal Protein method as documented in the Ideal Protein Clinic Manual and in the Ideal Protein Coaches Manual.
  Interventions: Behavioral: Ideal Protein Weight Loss Method
- Standard Weight Loss (Active Comparator): This arm utilizes evidence-based, low fat, low calorie strategies that have been shown to be effective for long-term weight loss and weight loss maintenance.
  Interventions: Behavioral: Standard Weight Loss

INTERVENTIONS:
Behavioral: Ideal Protein Weight Loss Method — An initial visit will take place in which each participant assigned to the experimental group will complete a health profile questionnaire.The Ideal Protein method will be explained and the participant will be weighed, measured and given diet related informational materials. A staff member will assist the participant with the selection of foods and snacks to ensure adequate quantity for the week. Weekly follow-up visits of 15 minutes duration will be implemented with a telephone follow-up occurring during the first 4 days after the initial appointment.
  For 12 weeks Ideal Protein foods that are of the appropriate composition and quantity will be provided at weekly or twice monthly intervals as included in the diet. Dietary supplements will be provided (multivitamin, calcium/magnesium, potassium, omega-3, and Ideal Salt substitute).
  Arms: Ideal Protein Weight Loss Protocol
Behavioral: Standard Weight Loss — This arm utilizes evidence-based strategies that have been shown to be effective for long-term weight loss and weight loss maintenance (including behavioral techniques, diet modification, and social support) consistent with the 2013 AHA/ACC/TOS Guideline for the Management of Overweight and Obesity in Adults. Participants in this arm will have an initial one hour consultation with a trained interventionist, where the fat goal and calorie restriction goal are explained.
  For 12 weeks low-fat reduced calorie foods that are of appropriate composition and quantity will be provided at weekly or twice monthly intervals as included in the diet. Dietary supplements will be provided (multivitamin, calcium/magnesium, potassium, omega-3, and Ideal Salt substitute).
  Arms: Standard Weight Loss

SUMMARY:
This study will examine whether, compared to a standard, low-fat, calorie-restricted diet intervention, the clinic-supported Ideal Protein weight loss method will result in greater weight loss and improvement in cardiometabolic risk factors over 3 months among obese adults with cardiovascular disease (CVD) risk factors.

DETAILED DESCRIPTION:
Restricting total calorie intake is emphasized in the 2013 American Heart Association/ American College of Cardiology/ The Obesity Society Guideline (AHA/ACC/TOS) for the Management of Overweight and Obesity in Adults for its effectiveness at reducing body weight and decreasing cardiometabolic risk factors. An implication of this focus on total quantity of calories consumed is that macronutrient composition of dietary intake and its effects on the hormonal milieu that regulates adipose accumulation in the human body do not play a significant role in weight loss. Such recommendations and the results of limited previous studies have led to the advice that all weight loss diets regardless of macronutrient composition will produce the same degree of weight loss if adherence to the diet is similar. In contrast, our previous studies have shown that despite comparable adherence to dietary goals, participants losing weight on a moderately carbohydrate-restricted, adequate protein regimen have improved cardiometabolic indicators as compared to those restricting fat. The RENEWAL trial will provide unique data on the efficacy of the Ideal Protein method (moderate carbohydrate restriction and adequate protein) for weight loss and improvement in cardiometabolic risk factors. The interventions will include a significant proportion of African-Americans, a group with very high rates of obesity which is often under-represented in trials examining the effects of weight loss diets. Findings from this trial may offer new evidence for the recommendation of specific macronutrient and behavioral approaches to the reduction of cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. All participants will be obese. Obesity will be defined as BMI ≥ 30 kg/m2 at the baseline study visit. An upper limit of BMI will be set at 49 kg/m2 to include a wide range of obese men and women with a reasonable probability of losing weight in the context of a dietary behavioral intervention.
2. Participants must have at least one co-morbid condition that increases risk of cardiovascular disease (history of CVD, type II diabetes mellitus, fasting plasma glucose>100 mg/dL, metabolic syndrome as defined by ATP III criteria, hypertension, hyperlipidemia, WC>40 in among men or >35 in among women).
3. All potential participants must be willing and able to provide informed consent.

Exclusion Criteria:

1. History of any bariatric surgery, including gastric banding, Roux-en-Y and duodenal switch with biliopancreatic diversion procedures, vertical banded gastroplasty, etc.
2. Currently on a diet or using prescription weight loss medications, and/or experienced weight loss >15 pounds within 6 months of study entry.
3. Regular use of alcohol >3 beverages per day or 21 beverages per week (1 standard beverage = 350 mL of 5% alcohol beer, or 150 mL of 12% wine, or 45 mL of 80-proof distilled spirits), amphetamines, cocaine, heroin, or marijuana over past 6 months.
4. Past or present history of eating disorder (including anorexia, bulimia or binge eating disorder) or severe/untreated psychiatric illness which may affect participation in study interventions.
5. Strict dietary concerns (e.g., vegetarian or kosher diet, significant nut or multiple food allergies). This is an exclusion because participant may not be able to fully participate in the intervention.
6. For women, current pregnancy or breastfeeding or plans to become pregnant during the study period. This is an exclusion because weight loss is contraindicated during pregnancy.
7. Plans to move out of the study area (>1 hour from study site) or difficulty to come to the study site. This is an exclusion because these conditions may interfere with the ability to fully participate in and complete the study.
8. Participation of another household member in the study; employees or persons living with employees of the study. This is an exclusion because randomization of more than one participant in a household to differing diets may cause conflict within a household and limit engagement in the intervention. Employees of the study are excluded due to potential conflicts of interest and knowledge of study assignments.
9. Participation in other lifestyle intervention trials currently. This is an exclusion because interference with ability to determine whether study interventions are responsible for outcomes.
10. Medical condition in which a carbohydrate restricted diet may not be advised (eg. severe renal impairment, osteoporosis, untreated thyroid disease, frequent gout attacks, Type I diabetes). This is an exclusion because participant may not be able to fully participate in the intervention.
11. Hospitalization for a CVD event such as myocardial infarction, stroke, TIA, coronary revascularization, heart failure, peripheral artery disease, or unstable angina within the last 6 weeks or unstable coronary artery disease. Major new medical illness including renal disease requiring dialysis, a life-threatening illness with life expectancy less than six months, or cancer requiring chemotherapy or radiation treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent.] This is an exclusion because these conditions may interfere with the ability to fully participate in and complete the study.
12. MMSE score < 23 or dementia. This is an exclusion because it may interfere with the ability to fully participate in the study.
13. Non-English speaking, a visual impairment or a hearing impairment that interferes with study participation. This is an exclusion criterion because these potential participants may not be able to participate fully in the intervention.
14. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in weight | Baseline and three months
  Change in weight at follow-up

SECONDARY OUTCOMES:
Body Composition | Baseline and three months
  Change in waist and hip circumference
Body Composition | Baseline and three months
  Change in lean and fat mass
Lipid parameters | Baseline and three months
  Change in lipid parameters
Fasting glucose | Baseline and three months
  Change in fasting glucose
Continuously measured glucose | Baseline and three months
  Change in continuously measured glucose
Systolic Blood Pressure | Baseline and three months
  Change in systolic blood pressure
Diastolic Blood Pressure | Baseline and three months
  Change in systolic blood pressure
Appetite | Baseline and three months
  Change in appetite as measured by self-report questionnaires
Satiety | Baseline and three months
  Change in satiety as measured by self-report questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Bogalusa Heart Study Clinic, Bogalusa, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fernandez CA, Potts K, Bazzano LA. Effect of ideal protein versus low-fat diet for weight loss: A randomized controlled trial. Obes Sci Pract. 2021 Oct 15;8(3):299-307. doi: 10.1002/osp4.567. eCollection 2022 Jun. PMID 35664249